CLINICAL TRIAL: NCT03257072
Title: Repeated Controlled Human Hookworm Infection in Healthy Dutch Volunteers
Brief Title: Repeated Controlled Human Hookworm Infection
Acronym: ReCHHI1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meta Roestenberg (Other)
Responsible Party: Sponsor-Investigator, Meta Roestenberg, Principal Investigator, Leiden University Medical Center
Organization: Leiden University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: ReCHHI1
Record Dates: First submitted 2017-08-10; First posted 2017-08-22 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Necator Americanus Infection
Keywords: hookworm; controlled human infection model
MeSH Terms: conditions — Ancylostomiasis

STUDY DESIGN:
Intervention Model Description: double-blind, placebo-controlled, dose-escalation trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A: 50 Necator americanus L3 larvae (Experimental): Mock infections with water at week 0 and 2, infection with 50 Necator americanus L3 larvae at week 4
  Interventions: Biological: 50 Necator americanus L3 larvae
- B: 100 Necator americanus L3 larvae (Experimental): Mock infections with water at week 0, infection with 50 Necator americanus L3 larvae at week 2 and 4
  Interventions: Biological: 100 Necator americanus L3 larvae
- C: 150 Necator americanus L3 larvae (Experimental): Infection with 50 Necator americanus L3 larvae at week 0, 2 and 4
  Interventions: Biological: 150 Necator americanus L3 larvae

INTERVENTIONS:
Biological: 50 Necator americanus L3 larvae — 1x50 Necator americanus L3 larvae
  Arms: A: 50 Necator americanus L3 larvae
Biological: 100 Necator americanus L3 larvae — 2x50 Necator americanus L3 larvae
  Arms: B: 100 Necator americanus L3 larvae
Biological: 150 Necator americanus L3 larvae — 3x50 Necator americanus L3 larvae
  Arms: C: 150 Necator americanus L3 larvae

SUMMARY:
Twenty-four healthy hookworm-naive volunteers will be exposed to 50 L3 Necator americanus larvae for a maximum of three times.

DETAILED DESCRIPTION:
Twenty-four volunteers will be allocated equally into three groups (i.e. group A, B, C). Group A, B, and C will have one, two, and three infections respectively. Every infection will be performed with 50 L3 Necator americanus larvae. Group A will receive infection at week 4 only. Group B will be infected at week 2 and week 4. Group C will be infected at week 0, 2 and 4. To maintain blinding, group A and B will receive mock infections with water at week 0 and week 0 and 2 respectively. The interval between each CHHI is 2 weeks. Before every infection, the safety will be assessed by a review of adverse events data with a local safety monitor.

Sixteen weeks after the last infection (week 20), all volunteers will be offered treatment with a 3-day regimen of albendazole to abrogate infection. Volunteers with average egg counts >250 eggs per gram will be asked if they would be willing to keep their infection for a maximum of two years (chronic donors). No more than four volunteers will be selected to be chronic donors. Six months after the last infection (or after the last donation for the chronic donors) volunteers will undergo their last visit.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is aged ≥ 18 and ≤ 45 years and in good health.
2. Subject has adequate understanding of the procedures of the study and agrees to abide strictly thereby.
3. Subject is able to communicate well with the investigator, is available to attend all study visits.
4. Subject agrees to refrain from blood donation to Sanquin or for other purposes throughout the study period.
5. For female subjects: subject agrees to use adequate contraception and not to breastfeed for the duration of study.
6. Subject has signed informed consent.

Exclusion Criteria:

1. Any history, or evidence at screening, of clinically significant symptoms, physical signs or abnormal laboratory values suggestive of systemic conditions, such as cardiovascular, pulmonary, renal, hepatic, neurological, dermatological, endocrine, malignant, haematological, infectious, immune-deficient, psychiatric and other disorders, which could compromise the health of the volunteer during the study or interfere with the interpretation of the study results. These include, but are not limited to, any of the following:

   * Body Mass Index (BMI) <18.0 or >30.0 kg/m2 at screening;
   * positive HIV, HBV or HCV screening tests;
   * the use of immune modifying drugs within three months prior to study onset (inhaled and topical corticosteroids and oral anti-histamines exempted) or expected use of such during the study period;
   * having one of the following laboratory abnormalities: ferritine <10 ug/L, transferrine <2.04 g/L or Hb <7.0 mmol/L for females or <8.0 mmol/L for males;
   * history of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years;
   * any history of treatment for severe psychiatric disease by a psychiatrist in the past year;
   * history of drug or alcohol abuse interfering with normal social function in the period of one year prior to study onset.
2. Known hypersensitivity to or contra-indications for use of albendazole, including co-medication known to interact with albendazole metabolism (e.g. carbamazepine, phenobarbital, phenytoin, cimetidine, theophylline, dexamethasone)
3. Known allergy to amphotericin B or gentamicin
4. For female subjects: positive urine pregnancy test at screening
5. Positive faecal qPCR or Kato-Katz for hookworm at screening, any known history of hookworm infection or treatment for hookworm infection or possible exposure to hookworm in the past
6. Being an employee or student of the department of parasitology of the LUMC
7. Current or past scars, tattoos, or other disruptions of skin integrity at the intended site of larval application
8. Subjects with planned travel to hookworm endemic areas during this trial
9. Receipt of a vaccine within 4 weeks prior to the study initiation
10. Known food allergy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events | 28 weeks
  Frequency of adverse events as compared between study groups A, B and C.
Magnitude of adverse events | 28 weeks
  Magnitude of adverse events as compared between study groups A, B and C.

SECONDARY OUTCOMES:
Variability in egg secretion | 20 weeks
  Variability in egg secretion by Kato-Katz from week 16 to 20
Lowest dose at which there is 100% patent hookworm infection | 20 weeks
  The lowest dose at which there is 100% patent hookworm infection, as defined by a positive Kato-Katz at any time between week 16 to 20
Comparison of the average number of eggs secreted | 20 weeks
  Comparison of the average number of eggs secreted by Kato-Katz and qPCR between different groups in weeks 16-20 after the infection

CONTACTS AND LOCATIONS:
Overall Officials: Meta Roestenberg, MD. PhD., Principal Investigator — LUMC
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hoogerwerf MA, Koopman JPR, Janse JJ, Langenberg MCC, van Schuijlenburg R, Kruize YCM, Brienen EAT, Manurung MD, Verbeek-Menken P, van der Beek MT, Westra IM, Meij P, Visser LG, van Lieshout L, de Vlas SJ, Yazdanbakhsh M, Coffeng LE, Roestenberg M. A Randomized Controlled Trial to Investigate Safety and Variability of Egg Excretion After Repeated Controlled Human Hookworm Infection. J Infect Dis. 2021 Mar 3;223(5):905-913. doi: 10.1093/infdis/jiaa414. PMID 32645714